CLINICAL TRIAL: NCT04385017
Title: Role of Inflammasomes in COVID-19 Disease
Acronym: CoVInnate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-PP-07
Record Dates: First submitted 2020-05-10; First posted 2020-05-12 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 by SARS-CoV-2 Infection

STUDY DESIGN:
Intervention Model Description: Patient with COVID-19 disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DNA from monocytes (Other): It will consist in the collection of 2 additional tubes at their blood draw. For DNA analysis, informed consent will be collected in writing
  Interventions: Other: COVID-19 patients

INTERVENTIONS:
Other: COVID-19 patients — It will consist in the collection of 2 additional tubes at their blood draw. For DNA analysis, informed consent will be collected in writing

SUMMARY:
As of March 25, 2020, 414,179 cases and 18,440 deaths secondary to Coronavirus 2019 disease (COVID-19) have been reported worldwide. The unfavorable course of the patients is characterized on the immunological level by an intense pro-inflammatory response which can go as far as a cytokinic storm. This pandemic affects a naive world population from an immunological point of view with respect to SARS-CoV-2 responsible for COVID-19. The evolution is favorable without hospitalization in almost 85% of cases. Among patients hospitalized for pneumonia, some will not require ventilatory support while others will need intensive care. To date, two main types of unfavorable evolution have been described. The first is a bi-phasic evolution beginning with a paucisymptomatic form which is worsened secondarily with respiratory distress associated with a decrease in the viral load in the airways. The second is associated with persistent high viral loads in the airways and detection of the virus in the blood. These different clinical profiles could depend on the quantitative and qualitative response of the innate immune system.

At the early stage of a viral infection the innate immunity is capable of detecting certain conserved microbial patterns (PAMP, pathogen-associated molecular pattern) recognized by receptors dedicated to these patterns (PRR, pattern recognition receptor). This process allows to initiate the pro-inflammatory response via different signaling pathways.

Activating multiprotein complexes called inflammasomes, which cause pro-IL-1β and pro-IL-18 to be transformed into active pro-inflammatory cytokines are one of these pathways.

The central role of inflammasomes in the secretion of these pro-inflammatory cytokines deserves an in-depth study of their activation during COVID-19, whereas the inadequate inflammatory response appears to be the determining factor in the unfavorable development of patients.

The objective of this project is to analyze the level of activation of the inflammasomes and then to search for inactivating or activating mutations among the genes which code for the proteins constituting the inflammasomes in Covid-19 patients. The identification of mutations in patients with a serious clinical presentation or even death would be followed by fundamental work by analyzing in a cellular model the impact of these mutations on the secretion of IL-1β.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old. SARS-CoV-2 infection confirmed by RT PCR or by serology Hospitalised patients with less than 14 days of COVID-19 symptoms. Date of first symptom being defined as to the date of one of the following symptoms : cough, dyspnea, fever above 38 °C, anosmia, dysgeusia or ageusia, chilblain Lupus erythematous Women of fertile age using at least one contraceptive method Health insurance Written informed consent

Exclusion criteria

* Pregnant or breastfeeding female
* Human immunodeficiency virus infection with CD4 under 200 cell/mm3
* Aplasia
* at-risk patients (minor, patient under judicial protection or tutorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Level of activation of inflammasomes in monocytes and polymorphonuclear neutrophils during COVID-19 | At inclusion
  Percentage of immune cells with inflammasome positive labeling using flow cytometry in comparison to controls

SECONDARY OUTCOMES:
Genes nucleoside polymorphism analysis | At inclusion
  Identification of genes nucleotide polymorphisms by Whole Exome Sequensing and bioinformatics analysis. Analysis of activating or inactivating mutations of NLRP3 NLRC4 AIM2 and Pyrin inflammasomes in patients with severe COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: COURJON Johan, Principal Investigator — CHU de Nice, Infectiologie
Locations (2):
- France (2):
  - Ch Cannes, Réanimation, Cannes, Alpes Maritimes
  - CHU de nice, Nice, Alpes-Maritimes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Courjon J, Dufies O, Robert A, Bailly L, Torre C, Chirio D, Contenti J, Vitale S, Loubatier C, Doye A, Pomares-Estran C, Gonfrier G, Lotte R, Munro P, Visvikis O, Dellamonica J, Giordanengo V, Carles M, Yvan-Charvet L, Ivanov S, Auberger P, Jacquel A, Boyer L. Heterogeneous NLRP3 inflammasome signature in circulating myeloid cells as a biomarker of COVID-19 severity. Blood Adv. 2021 Mar 9;5(5):1523-1534. doi: 10.1182/bloodadvances.2020003918. PMID 33683342